CLINICAL TRIAL: NCT01935531
Title: Prospective, Controlled and Monocentric Study to Evaluate the Effects of Topical 3% Diclofenac in 2.5% Hyaluronic Acid Gel on Tumor Metabolism in the Treatment of Actinic Keratoses in Immunocompetent and Immunocompromised Patients
Brief Title: Effects of Topical Diclofenac on Tumor Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Regensburg (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Professor Dr. Sigrid Karrer, Professor Dr., University Hospital Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Diclo-TuMet_01
Record Dates: First submitted 2013-08-30; First posted 2013-09-05 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Actinic Keratoses
Keywords: actinic keratoses; tumor metabolism; glycolysis; diclofenac; warburg effect
MeSH Terms: conditions — Keratosis, Actinic | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diclofenac (Experimental): 3 % diclofenac in 2.5% hyaluronic acid gel (Solaraze® 3% gel) is applied twice daily in the treatment area. 3 % diclofenac in 2.5% hyaluronic acid gel (Solaraze® 3% gel) is to be applied 1cm beyond the single AK.
  Interventions: Drug: 3% diclofenac in 2.5% hyaluronic acid gel

INTERVENTIONS:
Drug: 3% diclofenac in 2.5% hyaluronic acid gel
  Other Names: Solaraze Gel

SUMMARY:
The rationale of this study is to investigate the effects of topical diclofenac on tumor metabolism in the treatment of actinic keratoses in immunocompetent and immunocompromised patients.

Study hypothesis is that topical diclofenac lowers lactate level in skin biopsies of actinic keratoses. Planned number of patients is 38.

This study is a monocenter study investigating the effects of 3% diclofenac in 2.5% hyaluronic acid gel on tumor metabolism in the treatment of actinic keratoses. Treatment duration is 3 months. Skin biopsies will be obtained before treatment, at the end of the treatment and four weeks after the treatment. Control biopsies at visit 1 and 3 are performed in healthy, sun damaged and untreated skin. Evaluation of efficacy will be performed at the end of the treatment and four weeks after the treatment.

Duration of treatment is 3 months (±4 weeks). Approximately 0,5g Solaraze® 3% gel is applied on a 5cm x 5cm lesion. Solaraze® 3% gel is applied twice daily on the study lesions.

DETAILED DESCRIPTION:
Neoplastic cells show an increased glucose metabolism and glycolysis which is associated with high lactate concentrations. There is also data for several tumor entities that high levels of lactate in the tumor are associated with tumor progression, metastasis and poor clinical outcome. Kreutz et al. demonstrated that diclofenac inhibits tumor cell proliferation in vitro and tumor growth in vivo via COX-independent effects on glucose metabolism. Diclofenac is taken up by tumor cells and inhibits tumor cell proliferation through inhibition of the oncogene MYC and subsequently glycolysis and block of lactate transport. MYC regulates genes involved in glycolysis and is upregulated in neoplastic cells, which is in line with the metabolic switch to glycolysis, the so called "Warburg effect", that cancer cells show. Although these results were found in vitro using human melanoma cells and in vivo in a mouse model, a similar mechanism of action is assumed to be relevant for the treatment of actinic keratoses with topical diclofenac. However tumor metabolism in diclofenac-treated actinic keratoses has never been investigated. To investigate the mechanism of action of diclofenac in the treatment of actinic keratoses, a clinical study analyzing particularly lactate levels, glycolysis and inflammatory infiltrate is needed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been signed prior to or at Screening Visit
* Caucasian male and female patients
* Age > 18 years
* Negative pregnancy test in women of childbearing age
* Clinical diagnosis of actinic keratosis (AK)
* A minimum of three AK lesions

Exclusion Criteria in immunocompromised patients :

* Concomitant UV-phototherapy
* Pregnancy or lactation
* Women in child-bearing age who do not use highly efficient contraceptive methods (<1% failure rate per year)
* Skin diseases that might interfere with response evaluation of study treatment
* Topical pretreatment of the AK study lesions with photodynamic therapy, Solaraze® 3% gel, Aldara®, 5-FU, or polyphenon E during the 8 weeks preceding study treatment
* Radiation therapy performed in the treatment area during the 3 months preceding study therapy
* Systemic treatment with diclofenac
* Known intolerance to diclofenac or to any other ingredient of Solaraze® 3% gel
* Conditions that might interfere with the ability to understand the study and thus give written informed consent
* Simultaneous participation in another clinical study or participation in another clinical study in the 30 days directly preceding inclusion
* Suspected lack of compliance

Exclusion criteria in immunocompetent patients:

* Concomitant UV-phototherapy
* Pregnancy or lactation
* Women in child-bearing age who do not use highly efficient contraceptive methods (<1% failure rate per year)
* Patients with clinically relevant suppression of the immune system (e.g. drug induced, infection)
* Skin diseases that might interfere with response evaluation of study treatment
* Topical pretreatment of the AK study lesions with photodynamic therapy, Aldara®, Solaraze® 3% gel , 5-FU, or polyphenon E during the 8 weeks preceding study treatment
* Systemic treatment with cytostatic drugs or radiation therapy performed in the treatment area during the 3 months preceding study therapy
* Systemic treatment with diclofenac
* Known intolerance to diclofenac or to any other ingredient of Solaraze® 3% gel
* Conditions that might interfere with the ability to understand the study and thus give written informed consent
* Simultaneous participation in another clinical study or participation in another clinical study in participation in another clinical study in the 30 days directly preceding inclusion
* Suspected lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Lactate level in skin biopsies of actinic keratoses | 4 weeks after the treatment
  Assessment of the effects of topical 3% diclofenac in 2.5% hyaluronic acid gel on lactate level in skin biopsies of actinic keratoses. Skin biopsies of actinic keratoses are obtained prior to treatment and 4 weeks after the treatment.

SECONDARY OUTCOMES:
Lactate level in skin biopsies of healthy skin in a subpopulation | Before treatment and 4 weeks after the treatment
  Assessment of the effects of topical 3% diclofenac in 2.5% hyaluronic acid gel on lactate level in skin biopsies of actinic keratoses compared to untreated sun damaged, healthy skin in a subpopulation
Glycolysis-relevant proteins evaluated using PCR and Westernblot techniques | at the end of the treatment and 4 weeks after the treatment
  Glycolysis-relevant proteins evaluated using PCR and Westernblot techniques
Metabolic changes (e.g. glucose, amino acids) | at the end of the tretment and 4 weeks after the treatment
  Metabolic changes (e.g. glucose, amino acids) evaluated by NMR methods and bioluminescence imaging techniques

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Regensburg, Regensburg, Bavaria, Germany

REFERENCES:
- [Derived] Singer K, Dettmer K, Unger P, Schonhammer G, Renner K, Peter K, Siska PJ, Berneburg M, Herr W, Oefner PJ, Karrer S, Kreutz M, Datz E. Topical Diclofenac Reprograms Metabolism and Immune Cell Infiltration in Actinic Keratosis. Front Oncol. 2019 Jul 3;9:605. doi: 10.3389/fonc.2019.00605. eCollection 2019. PMID 31334125